CLINICAL TRIAL: NCT03381495
Title: The Association Between Epidural Labor Analgesia and Pregnancy Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deng Dongrui (Other)
Responsible Party: Sponsor-Investigator, Deng Dongrui, professor,chief doctor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-C20171201
Record Dates: First submitted 2017-12-02; First posted 2017-12-22 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Labor Pain; Pregnancy Outcomes; Psychological Disorder
Keywords: Epidural Labor Analgesia; length of labor stage; fetal outcomes; maternal outcomes; postpartum depression; exercise
MeSH Terms: conditions — Labor Pain; Mental Disorders; Depression, Postpartum; Motor Activity | interventions — Ropivacaine; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural analgesia during labor (Experimental): The epidural analgesia technique was used to maintain analgesia for parturients who request labor analgesia.First, we injected a test dose of 5ml 1% lidocaine . If not adverse effects were observed 10 minutes after the test dose, the parturient then received a bolus injection of an initial dose of 8-10 ml mixed liquids of 0.075% ropivacaine and 0.2ug/ml sufentanil citrate. We then connected the epidural catheter with a patient-controlled epidural analgesia (PCA) pump, which provided patients the same mixed solution at 8-10ml/h until the delivery of neonates.
  Interventions: Drug: Ropivacaine Hydrochloride, Sufentanil
- Non-epidural analgesia during labor (No Intervention): Women who refused epidural labor analgesia were included in the non-epidural analgesia group, and they don't receive epidural analgesia during labor

INTERVENTIONS:
Drug: Ropivacaine Hydrochloride, Sufentanil — In this research one group will receive epidural analgesia(Ropivacaine Hydrochloride, Sufentanil), data will be collected and analyzed between this group and non-epidural analgesia group.
  Arms: Epidural analgesia during labor

SUMMARY:
Labor analgesia can alleviate intrapartum pain, in the importance of the delivery is very obvious.But some researches think labor analgesia may affect the progress of labor, increase the cesarean section rate.This research adopts the epidural anesthesia to study labor analgesia effects on delivery outcomes and long-term emotional and psychological effects on the mothers. Besides, we also want to study the effect of exercise during pregnancy on the mode of delivery.

ELIGIBILITY:
Inclusion Criteria:

healthy and full term pregnant women

Exclusion Criteria:

the pregnant women with complications

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Labor duration | At the end of the delivery
  Duration of three stages of labor.

SECONDARY OUTCOMES:
1 minute Apgar index | 1 minute after the infant is born
  The index indicates the infant s' conditions, including heart rate, breathing, muscle tone, reflex response, color. Each characteristic is given an individual score; two points for each of the five categories if all is completely well; then all scores are totaled. The score is from 0 to 10.
5 minute Apgar index | 5 minutes after the infant is born
  The index indicates the infant s' conditions, including heart rate, breathing, muscle tone, reflex response, color. Each characteristic is given an individual score; two points for each of the five categories if all is completely well; then all scores are totaled. The score is from 0 to 10.
Visual Analogue Scores(VAS) | 5min before analgesia;5min,15min, 30min,60min after analgesia; at the time of latent phase, active phase, full dilation of the cervix, crowning of head, and laceration repair.
  VAS is the most common pain scale for quantification. The score is from 0 to 10. The score is higher, the patient will be more painful. That will indicate if the analgesia is effective.
Modified Bromage scores | 5min before analgesia;5min,15min, 30min,60min after analgesia; at the time of latent phase, active phase, full dilation of the cervix, crowning of head, and laceration repair.
  The modified Bromage score is the most frequently used measure of motor block. The scores is from 0 to 3. In this scale, the intensity of motor block is assessed by the patient's ability to move their lower extremities (0: no motor paralysis; 1: inability to raise extended leg, but able to move knee and foot; 2: inability to raise extended leg and to move knee, but able to move foot; 3: inability to raise extended leg or to move knee and foot). That will indicate if the analgesia block the patient motor too much.
Postpartum depression | 3 days after delivery,6 weeks after delivery, 3 months after delivery, 6 months after delivery, 1 year after delivery.
  Assess the risk of postpartum depression among all participants using EPDS，HAMA.
The mode of delivery | At the end of delivery
  Including spontaneous vaginal delivery, vacuum- and forceps-assisted delivery, cesarean delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zha Y, Gong X, Yang C, Deng D, Feng L, Luo A, Wan L, Qiao F, Zeng W, Chen S, Wu Y, Han D, Liu H. Epidural analgesia during labor and its optimal initiation time-points: A real-world study on 400 Chinese nulliparas. Medicine (Baltimore). 2021 Mar 5;100(9):e24923. doi: 10.1097/MD.0000000000024923. PMID 33655955